CLINICAL TRIAL: NCT06812494
Title: A Randomized, Double Blind, Controlled, Phase 2 Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Neutralization of VRC07-523LS, PGT121.414.LS, and PGDM1400LS Broadly Neutralizing Monoclonal Antibodies Given Intravenously in Adult Participants Without HIV
Brief Title: A Study of VRC07-523LS, PGT121.414.LS, and PGDM1400LS Broadly Neutralizing Monoclonal Antibodies Given Intravenously in Adult Participants Without HIV
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH); Department of Health and Human Services (U.S. Federal Agency); Dale and Betty Bumpers Vaccine Research Center (VRC) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 206/HPTN 114; 39137 (Other: DAIDS-ES ID)
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: HIV
Keywords: HIV Prevention; bnAb; Monoclonal antibody; Intravenous; Triple combination; VRC07-523LS; PGT121.414.LS; PGDM1400LS

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (400 mg + 400 mg +400 mg) (Experimental): VRC07-523LS 400mg + PGT121.414.LS 400mg + PGDM1400LS 400mg to be administered via IV infusion sequentially in this order at Month 0 and Month 6
  Interventions: Biological: VRC07-523LS 400mg; Biological: PGT121.414.LS 400mg; Biological: PGDM1400LS 400mg
- Group 2 (3200 mg + 1600 mg +1600 mg) (Experimental): VRC07-523LS 3200mg + PGT121.414.LS 1600mg + PGDM1400LS 1600mg to be administered via IV infusion sequentially in this order at Month 0 and Month 6
  Interventions: Biological: VRC07-523LS 3200mg; Biological: PGT121.414.LS 1600mg; Biological: PGDM1400LS 1600mg

INTERVENTIONS:
Biological: VRC07-523LS 400mg — Intravenous infusion (IV)
  Arms: Group 1 (400 mg + 400 mg +400 mg)
Biological: PGT121.414.LS 400mg — IV infusion
  Arms: Group 1 (400 mg + 400 mg +400 mg)
Biological: PGDM1400LS 400mg — IV infusion
  Arms: Group 1 (400 mg + 400 mg +400 mg)
Biological: VRC07-523LS 3200mg — IV infusion
  Arms: Group 2 (3200 mg + 1600 mg +1600 mg)
Biological: PGT121.414.LS 1600mg — IV infusion
  Arms: Group 2 (3200 mg + 1600 mg +1600 mg)
Biological: PGDM1400LS 1600mg — IV infusion
  Arms: Group 2 (3200 mg + 1600 mg +1600 mg)

SUMMARY:
HVTN 206/HPTN 114 is a randomized, double blind, controlled, phase 2 clinical trial to evaluate the safety, tolerability, pharmacokinetics, and neutralization of VRC07-523LS, PGT121.414.LS, and PGDM1400LS broadly neutralizing monoclonal antibodies given intravenously in adult participants without HIV.

The hypothesis of the study is that the combination of VRC07-523LS and PGT121.414.LS and PGDM1400LS antibodies when administered via the intravenous (IV) route will be safe and tolerable in adult participants without HIV.

The study aims to enroll 200 participants across multiple sites with an estimated total duration of participation of eighteen (18) months.

ELIGIBILITY:
Inclusion Criteria:

* Participants need to be between 18 and 65 years old.
* Participants must have access to a participating clinical research site and be willing to follow the study schedule.
* Participants should understand the study details and be willing to give informed consent.
* Participants must agree not to join any other clinical trials until they finish this study.
* Participants must be willing to receive HIV test results.
* Participants should be open to discussing HIV prevention.
* Clinic staff should assess participants as having a low risk of getting HIV, and participants must commit to avoiding high-risk behaviors during the study.
* Hemoglobin: Participant meets minimum levels depending on gender and hormone therapy status.
* White Blood Cells (WBC): Should be within the normal range or approved by a site clinician.
* Platelets: At least 100,000 cells/mm³.
* Alanine aminotransferase (ALT): Less than 5 times the upper normal limit.
* Creatinine: Less than 1.8 times the upper normal limit or less than 1.5 times your baseline level.
* Participants must test negative for HIV-1 and HIV-2.
* Participants urine protein must be negative or trace.

Reproductive Status:

* Participants of child-bearing potential need a negative pregnancy test within 72 hours before starting the study.
* Participants must agree to use effective birth control from at least 21 days before joining the study until the end of the study.
* Participants must agree not to try to become pregnant through any method during the study.

Exclusion Criteria:

* Participants cannot have had a blood transfusion within the last 120 days.
* Participants cannot have received experimental treatments within the last 30 days.
* Participants cannot weigh less than 35 kg (about 77 lbs).
* Participants cannot plan to join another clinical trial during this study.
* Participants cannot be pregnant or breastfeeding.
* Participants cannot have received an HIV vaccine in a previous trial (unless it was a placebo, subject to Protocol Safety Review Team's approval).
* Participants cannot have had any live vaccines within the last 14 days or non-live vaccines within the last 7 days.
* Participants cannot have had humanized or human monoclonal antibodies recently, except for certain HIV antibodies more than 12 months ago.
* Participants cannot have had allergy shots within the last 14 days.
* Participants cannot have taken immunosuppressive drugs within the last 30 days, with some exceptions like nasal sprays or mild skin treatments.
* Participants cannot participate if they have had serious allergic reactions to the components of the study product.
* Participants cannot have received immunoglobulin within the last 60 days.
* Participants cannot have an autoimmune disease that requires immunosuppressive treatment, unless it's mild and stable.
* Participants cannot have an immune system deficiency.
* Participants cannot have any significant medical condition or abnormal lab results that could impact their health during the study.
* Participants cannot have conditions that make repeated injections or blood draws difficult.
* Participants cannot have conditions requiring active medical treatment that could pose a risk during the study.
* Participants cannot have conditions that could be confused with reactions to the study product.
* Participants cannot have medical, social, or occupational conditions that would interfere with the study.
* Participants cannot have severe psychiatric conditions, like ongoing risk of suicide or recent history of suicide attempts.
* Participants cannot be undergoing treatment for tuberculosis.
* Participants cannot have severe asthma that requires frequent medication or emergency care.
* Participants cannot have diabetes mellitus (DM) (well-controlled Type 2 DM or an isolated history of gestational diabetes are not exclusionary).
* Participants blood pressure must be below 160/110 mmHg.
* Participants cannot have any diagnosed bleeding disorders.
* Participants cannot have active cancer but may be eligible if, in the investigator's estimation, they have a reasonable assurance of sustained cure, or are unlikely to experience recurrence of malignancy during the period of the study
* Participants cannot have had seizures or taken seizure medications in the past 3 years.
* Participants cannot have a history of severe allergic reactions like anaphylaxis, unless it has been well-controlled for at least 5 years.
* Participants cannot have acute or unstable hepatitis B or C, but stable chronic cases may be considered.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing local Adverse Events (AEs) | At Days 1, 4, 7, 169 and 173
Percentage of participants experiencing local AEs | At Days 1, 4, 7, 169 and 173
Number of participants experiencing systemic AEs | At Days 1, 4, 7, 169 and 173
Percentage of participants experiencing systemic AEs | At Days 1, 4, 7, 169 and 173
Number of participants experiencing unsolicited AEs | Baseline through Week 48
Percentage of participants experiencing unsolicited AEs | Baseline through Week 48
Number of participants experiencing Serious Adverse Events | Baseline through Week 48
Number of participants who discontinue study product administration and terminate the study early | Baseline through Week 48
Percentage of participants who discontinue study product administration and terminate the study early | Baseline through Week 48
Change from baseline in ALT | Baseline, Days 1, 57, 169, 225 and 337
Change from baseline in aspartate aminotransferase (AST) | Baseline, Days 1, 57, 169, 225 and 337
Change from baseline in alkaline phosphatase (Alk Phos) | Baseline, Days 1, 57, 169, 225 and 337
Change from baseline in creatinine | Baseline, Days 1, 57, 169, 225 and 337
Change from baseline in Complete Blood Count (CBC) | Baseline, Days 1, 57, 169, 225 and 337

SECONDARY OUTCOMES:
Area under the curve (AUC) of VRC07-523LS, PGDM1400LS, and PGT121.414.LS | At Days 1, 4, 7, 29, 57, 169, 225 and 337
Maximum concentration (C(max)) of VRC07-523LS, PGDM1400LS, and PGT121.414.LS | At Days 1, 4, 7, 29, 57, 169, 225 and 337
Time to C(max) (T(max)) of VRC07-523LS, PGDM1400LS, and PGT121.414.LS | At Days 1, 4, 7, 29, 57, 169, 225 and 337
Clearance (CL) of VRC07-523LS, PGDM1400LS, and PGT121.414.LS | At Days 1, 4, 7, 29, 57, 169, 225 and 337
Volume of distribution (Vd) of VRC07-523LS, PGDM1400LS, and PGT121.414.LS | At Days 1, 4, 7, 29, 57, 169, 225 and 337
Terminal elimination rate constant (λz) of VRC07-523LS, PGDM1400LS, and PGT121.414.LS | At Days 1, 4, 7, 29, 57, 169, 225 and 337
Terminal half-life (T1/2) of VRC07-523LS, PGDM1400LS, and PGT121.414.LS | At Days 1, 4, 7, 29, 57, 169, 225 and 337
Area under the magnitude-breadth curve (AUC-MB) of VRC07-523LS, PGDM1400LS, and PGT121.414.LS | At Days 1, 4, 7, 29, 57, 169, 225 and 337
Presence of antidrug antibodies (ADAs) for VRC07-523LS, PGDM1400LS, and PGT121.414.LS | At Days 1, 169 and 337

CONTACTS AND LOCATIONS:
Locations (21):
- United States (13):
  - Alabama CRA (Site #31788), Birmingham, Alabama
  - Bridge HIV, San Francisco Department of Public Health, San Francisco, California
  - The Hope Clinic of the Emory Vaccine Research Center; Emory University, Decatur, Georgia
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Fenway Health, Boston, Massachusetts
  - BIDMC VCRS (Site ID# 32077), Boston, Massachusetts
  - Columbia P&S CRS, New York, New York
  - University of Rochester Vaccines to Prevent HIV Infection CRS (Site ID 31467), Rochester, New York
  - Chapel Hill CRS (Site #3201), Chapel Hill, North Carolina
  - Penn Prevention CRS, Philadelphia, Pennsylvania
  - University of Pittsburgh CRS (Site 1001), Pittsburgh, Pennsylvania
  - Vanderbilt Vaccine (VV) CRS, Nashville, Tennessee
  - Seattle Vaccine and Prevention CRS (Site ID# 30331), Seattle, Washington
- Instituto de Pesquisa Clinica Evandro Chagas (IPEC) CRS, Rio de Janeiro, Brazil
- Peru (3):
  - ACSA CRS, Iquitos, Maynas
  - CITBM CRS (Site ID 31970), Callao
  - Via Libre (Site ID 31909), Lima
- South Africa (4):
  - Perinatal HIV Research Unit (PHRU), Johannesburg, Gaunteng
  - Chatsworth CRS, Chatsworth, KwaZulu-Natal
  - Setshaba Research Centre, Soshanguve-H, Soshanguve
  - Groote Schuur HIV CRS, Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.hptn.org/research/studies/hvtn-206hptn-114